CLINICAL TRIAL: NCT03177252
Title: Scalp Block: Hemodynamic Stability and Patient Comfort In Craniotomy Patients
Acronym: Scalp block
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator decided not to go forward with the trial.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201701037
Record Dates: First submitted 2017-05-08; First posted 2017-06-06 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Tumor, Brain; Anesthesia, Local
MeSH Terms: conditions — Brain Neoplasms | interventions — Lidocaine; Sodium Chloride; Saline Solution; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Scalp block with lidocaine and bupivacaine (Experimental): * Scalp block with a mixture of 2% lidocaine and 0.5% bupivacaine
  * Once the surgery is completed, patients will be awaken and extubated following a basic neurological exam. If the extubation is delayed or if the patient is taken to ICU intubated, those patients will be excluded from the study.
  Interventions: Drug: Lidocaine; Drug: Bupivacaine
- Scalp block with saline (Placebo Comparator): * Scalp block with saline
  * Once the surgery is completed, patients will be awaken and extubated following a basic neurological exam. If the extubation is delayed or if the patient is taken to ICU intubated, those patients will be excluded from the study.
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Lidocaine — -2% lidocaine will be given
  Arms: Scalp block with lidocaine and bupivacaine
Drug: Sodium chloride — -Normal saline will be given
  Other Names: Saline; Normal Saline
  Arms: Scalp block with saline
Drug: Bupivacaine — -0.5% bupivacaine will be given
  Arms: Scalp block with lidocaine and bupivacaine

SUMMARY:
Making sure the heart rate and or the blood pressure [called hemodynamic instability] during surgery is stable, setting up for a rapid postoperative recovery, and ensuring that patients have adequate pain relief are some of the important goals of neurosurgical anesthesia. Scalp block anesthesia [injection of a numbing agent into the area of the scalp where the incision will be] together with general anesthesia is used to achieve these goals. There has been some research on whether or not scalp block improves patient recovery and pain management, but the studies have not be large enough to say for certain. This is true even though scalp block is used with almost every patient that is having brain surgery. The investigators propose to determine if scalp block in combination with asleep anesthesia is better than asleep anesthesia alone in patients who are having brain surgery for tumors in the cerebral area of the brain.

DETAILED DESCRIPTION:
Avoidance of hemodynamic fluctuations in the heart rate and or the blood pressure perioperatively, rapid postoperative recovery, and adequate postoperative pain relief are some of the important goals of neurosurgical anesthesia. Scalp block in association with general anesthesia is used to achieve these goals. Previous studies have been published related to the effect of scalp block on the perioperative outcomes on the craniotomy patients. The results reported so far are controversial and one cannot at this point define a positive effect for post-operative pain relief. This disparity in results may be the consequences of the size of the patient population. However scalp block is an accepted practice in the craniotomy patients. The investigators believe this is the first study which assesses the effectiveness of scalp block for asleep craniotomy with the largest sample size study so far conducted in the literature related to this topic. The aim of this study is to assess the effectiveness of scalp block for the perioperative comfort of the craniotomy patients undergoing resection for supratentorial tumors.

After the consent for the participation and enrollment in the study is done, patients will be randomized to two groups, a study group will receive a scalp block with a mixture of 2% lidocaine and 0.5% bupivacaine while the control group will receive the scalp block with saline. Intraoperatively, all patients will be preoxygenated, fentanyl (1-2mcg/kg) will be given and anesthesia will be induced with propofol (1-2mg/kg) and lidocaine (1-1.5mg/kg). Tracheal intubation will be facilitated by using either rocuronium (0.6 mg/kg) or succinylcholine (1-1.5mg/kg) intravenously. The lungs will be ventilated with a fresh gas flow of oxygen for 2 minutes before tracheal intubation with cuffed oral endotracheal tube. Anesthesia will be maintained with inhalational anesthetic Isoflurane, Sevoflurane or Desflurane (0.8-1 MAC) and fentanyl infusion (1-2mcg/kg) with the dose adjusted according to the patient's hemodynamics. Bilateral BIS or EEG to maintain an adequate level of depth of anesthesia will be used whenever feasible. After intubation, a scalp block will be performed. The randomization of the scalp block syringes will be provided by the pharmacy and neither the scalp block performer nor the attending will be aware of the syringe content. To standardize the block, a pain specialist is involved. Response to the pinning will be assessed using the hemodynamic parameters and rescue analgesics (fentanyl bolus 50 - 100 mcg) and/or propofol bolus 50 - 100 mg will be given as a bolus if significant response is noted. Significant response being a rise in the patient's heart rate and/or the blood pressure more than 20% from the patient's baseline heart rate and/or the blood pressure just before pinning. Similarly, response to the surgical incision will be noted and rescue analgesics will be given if needed. Intraoperative propofol requirement and opioid requirements will be recorded. The post-operative orders for pain control will be standardized for all the patients.

ELIGIBILITY:
Inclusion Criteria:

->18years of age undergoing elective craniotomy for supratentorial tumors

Exclusion Criteria:

* Age group < 18
* Emergency craniotomies
* Infratentorial tumors.
* Patients who need intraoperative evoked potential monitoring which precludes the scalp block.
* Patients with known cranial defects.
* Patients who are on medications for chronic pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall perioperative comfort of the patient as measured by hemodynamic fluctuations | Up to 48 hours
  Hemodynamic fluctuations during pinning of the head with a Mayfield head-holder and skin incision which represents the most extreme painful stimulation for the entire surgery (significant response being rise in the patient's heart rate and/or the blood pressure more than 20% from the patient's baseline heart rate and/or the blood pressure prior pinning)
Overall perioperative comfort as measured by opioid requirements | Up to 48 hours
  Overall perioperative opioid requirements until the next morning of the surgery as an overall evaluation of the patient's comfort.

SECONDARY OUTCOMES:
Cost-effectiveness of scalp block | Up to 48 hours
  Scalp block for the craniotomy
  1. lowers overall administration of opioids, which will decrease the side effects of opioids
  2. improve the immediate postoperative pain which may decrease the occurrence of chronic postoperative pain and
  3. may result in the early discharge from the hospital contributing to shorter hospital stay reducing the financial burden for both the patient and the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Umeshkumar Athiraman, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu